CLINICAL TRIAL: NCT00275041
Title: Phase II Trial of Concurrent Irinotecan Plus Cetuximab in Patients With Advanced Breast Cancer With Prior Anthracycline and/or Taxane-Containing Therapy
Brief Title: Irinotecan and Cetuximab in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0436; NCI-2012-02679 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000456255 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Cetuximab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cetuximab + irinotecan (Experimental): Patients receive cetuximab IV over 1-2 hours on days 1, 8, and 15 and irinotecan hydrochloride IV over 1½ hours on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  After completion of study treatment, patients are followed periodically for up to 5 years.
  Interventions: Biological: cetuximab; Drug: irinotecan hydrochloride

INTERVENTIONS:
Biological: cetuximab
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving irinotecan together with cetuximab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving irinotecan together with cetuximab works in treating patients with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the antitumor activity, by confirmed response rate, of concurrent irinotecan hydrochloride and cetuximab in patients with metastatic breast cancer with prior anthracycline and/or taxane-containing therapy.

Secondary

* Estimate 6-month, progression-free survival of patients.
* Evaluate the adverse event profile of irinotecan hydrochloride in combination with cetuximab in patients with metastatic breast cancer.
* Estimate progression-free survival of patients.
* Estimate overall survival.

OUTLINE: Patients receive cetuximab IV over 1-2 hours on days 1, 8, and 15 and irinotecan hydrochloride IV over 1½ hours on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 5 years.

PROJECTED ACCRUAL: A total of 38 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast

  * Clinical manifestations of metastatic disease
* If patient's tumor is HER2 positive (3+ by immunohistochemistry [IHC] or amplified by fluorescent in situ hybridization [FISH]), must have received at least one prior trastuzumab (Herceptin)-containing regimen unless there is a contraindication
* Measurable disease defined as at least one lesion whose longest diameter can be accurately measured

  * The only evidence of metastasis must not be bone metastases or other non-measurable disease
  * Nonmeasurable disease is defined as all other lesions, including small lesions (longest diameter < 2 cm) and truly nonmeasurable lesions which include any of the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Cystic lesions
    * Abdominal masses that are not confirmed and followed by imaging techniques
* No known CNS metastasis unless controlled by prior surgery and/or radiotherapy

  * To be considered controlled, there must be at least 2 months of no symptoms or evidence of progression prior to study entry
* Hormone receptor status

  * Not specified

PATIENT CHARACTERISTICS:

* Men or women
* Menopausal status not specified
* ECOG performance status 0-2
* Life expectancy > 3 months
* Hemoglobin > 8.0 g/dL
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin normal
* AST and ALT ≤ 5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must employ adequate contraception (as determined by the treating physician) during treatment and for 30 days after treatment ends
* Disease-free for ≥ 3 years of other invasive non-breast malignancies (exception: curatively treated basal cell or squamous cell carcinoma of the skin and carcinoma in situ of the cervix)
* No history of allergy or hypersensitivity to drug product excipients, murine antibodies, or agents chemically similar to irinotecan and/or cetuximab
* No history or evidence of Gilbert's syndrome
* No active, unresolved infection
* No New York Heart Association class III or IV cardiovascular disease
* No serious concomitant medical condition that would make it undesirable for patient to participate in the trial or would jeopardize compliance with protocol treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No more than 2 prior chemotherapy regimens in the metastatic setting (irrespective of hormonal therapy or prior trastuzumab therapy)

  * Prior treatment in the metastatic or adjuvant setting must have included an anthracycline or a taxane
* No major surgery ≤ 3 weeks prior to registration
* No chemotherapy ≤ 2 weeks prior to registration
* No radiotherapy ≤ 4 weeks prior to registration
* No prior irinotecan hydrochloride
* No prior therapy with an epidermal growth factor receptor (EGFR) antagonist (either monoclonal antibody or tyrosine kinase inhibitor), such as gefitinib or erlotinib
* No prior therapy with a dual EGFR/HER2 inhibitor (e.g., lapatinib)
* No concurrent interleukin-11(oprelvekin)
* Routine use of granulocyte colony stimulating factors (CSFs) is not permitted during course 1 of this study

  * Subsequent use of CSFs is permitted at the discretion of the treating investigator
* No other concurrent antitumor therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-02; Primary Completion 2007-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Confirmed tumor response (complete or partial) | Up to 5 years

SECONDARY OUTCOMES:
Time to disease progression | Up to 5 years
Survival time | Up to 5 years
Progression-free survival at 6 months | at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Hobday, MD, Study Chair — Mayo Clinic

REFERENCES:
- [Background] Reinholz MM, Kitzmann KA, Tenner K, Hillman D, Dueck AC, Hobday TJ, Northfelt DW, Moreno-Aspitia A, Roy V, LaPlant B, Allred JB, Stella PJ, Lingle WL, Perez EA. Cytokeratin-19 and mammaglobin gene expression in circulating tumor cells from metastatic breast cancer patients enrolled in North Central Cancer Treatment Group trials, N0234/336/436/437. Clin Cancer Res. 2011 Nov 15;17(22):7183-93. doi: 10.1158/1078-0432.CCR-11-0981. Epub 2011 Oct 5. PMID 21976532
- [Background] Reinholz MM, Kitzmann KA, Hobday TJ, et al.: Cytokeratin-19 (CK19) and mammaglobin (MGB1) gene expression in circulating tumor cells (CTCs) from metastatic breast cancer patients enrolled in the NCCTG trials, N0436 and N0437. [Abstract] J Clin Oncol 27 (Suppl 15): A-11095, 2009.